CLINICAL TRIAL: NCT04003350
Title: The Effect of Prolonged Multimodal Analgesic Regimen on Post Hospital Discharge Opioid Use and Pain Control After Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019MAUSTKA
Record Dates: First submitted 2019-06-21; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Oxycodone; Tramadol; Acetaminophen; Meloxicam; Gabapentin; metaxalone; Esomeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Regimen (Active Comparator): Weeks 1-4
  * Oxycodone 5 mg PRN q4h (30 tablets)
  * Tramadol 50 mg PRN q6h (30 tablets)
  Interventions: Drug: Oxycodone; Drug: Tramadol
- Multimodal pain regimen with PRN opioids (Experimental): Weeks 1-4
  * Tylenol 1000 mg q8h (standing)
  * Meloxicam 15 mg qD (standing).
  * Gabapentin 200 mg BID (with morning and evening Tylenol dose)
  * Metaxalone 800mg PO TID (Tizanidine 2mg q8h if insurance coverage is not possible for metaxalone)
  * Esomeprazole 20mg daily if not already on another H2 blocker or PPI
  * Oxycodone 5 mg PRN q4h (30 tablets)
  * Tramadol 50 mg PRN q6h (30 tablets)
  Interventions: Drug: Oxycodone; Drug: Tramadol; Drug: Tylenol; Drug: Meloxicam; Drug: Gabapentin; Drug: Metaxalone; Drug: Esomeprazole 20mg

INTERVENTIONS:
Drug: Oxycodone — Patients are given, for up to 4 weeks, Oxycodone 5m PRN every four hours (up to 30 tablets)
Drug: Tramadol — Patients are given, for up to 4 weeks, Tramadol 50mg PRN every 6 hours (up to 30 tablets)
Drug: Tylenol — Tylenol 1000 mg: take as needed every 8 hours
  Arms: Multimodal pain regimen with PRN opioids
Drug: Meloxicam — Meloxicam 15 mg as need once per day
  Arms: Multimodal pain regimen with PRN opioids
Drug: Gabapentin — •Gabapentin 200 mg with morning and evening Tylenol dose
  Arms: Multimodal pain regimen with PRN opioids
Drug: Metaxalone — Metaxalone 800mg TID
  Arms: Multimodal pain regimen with PRN opioids
Drug: Esomeprazole 20mg — Esomeprazole 20mg daily
  Arms: Multimodal pain regimen with PRN opioids

SUMMARY:
It is well recognized that a multimodal analgesia program targeting multiple pain pathways, is more effective for controlling pain during the hospital stay and in the acute postoperative period than monotherapy-based regimens, such as opioids only. This multimodal analgesic regimen also leads to reduce opioid consumption and its related side effects after hip and knee joint replacement procedures. One potential strategy to reduce the use of opioids after TKA is to administer a prolonged oral multimodal pain regimen that targets multiple pain pathways in the post hospital discharge period. This can be equal or more effective than the regimen of opioid prescriptions used after TKA. To the best of our knowledge, there have been no studies conducted that directly examine the effect of prolonged multimodal pain regimen after hospital discharge in primary TKA patients.

PURPOSE:

1. To determine whether a prolonged multimodal pain regimen after discharge from primary TKA can provide equivalent or better pain control while reducing opioid consumption and, subsequently, opioid-related side effects.
2. To determine whether patient expectations and routine opioid prescription practices at the time of discharge from primary TKA impacts opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary TKA with underlying diagnosis of osteoarthritis.
* ASA I - III
* Spinal anesthesia
* All patients will have cemented total knee utilizing a medial parapatellar approach including patellar resurfacing. A tourniquet will be used in all cases
* Male and Female over 18 who are willing and able to provide informed consent

Exclusion Criteria:

* Opioid use within 3 months preoperatively
* Inability to take the protocol medications
* Anticoagulant other than aspirin
* Contraindication to regional anesthesia
* Non-english speaking
* ASA IV or greater
* Psychiatric or cognitive disorders
* Allergy/contraindications to protocol medications.
* Renal insufficiency with Cr > 2.0 or hepatic failure
* General anesthesia
* Sensory/motor disorder involving the operative limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | Postsurgery days 1-30
  Measured via Visual Analog scale (0-100mm)
Opioid related side effects | post-surgery days 1-30
  Severity measured via Visual Analog scale (0-100mm)

SECONDARY OUTCOMES:
opioid consumption | post-surgery weeks 1-4
  morphine milligram equivalent
opioid consumption | post-surgery weeks 1-4
  number of pills consumed
number of opioid refills | post-surgery weeks 1-4
  number of times subjects asked to have an opioid prescription refilled during post-operative period
90 day complications | post-surgery 90 days
  collection of all post-operative medical complications within the first 90 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Li WT, Bell KL, Yayac M, Barmann JA, Star AM, Austin MS. A Postdischarge Multimodal Pain Management Cocktail Following Total Knee Arthroplasty Reduces Opioid Consumption in the 30-Day Postoperative Period: A Group-Randomized Trial. J Arthroplasty. 2021 Jan;36(1):164-172.e2. doi: 10.1016/j.arth.2020.07.060. Epub 2020 Jul 30. PMID 33036845